CLINICAL TRIAL: NCT05102942
Title: A Randomized Controlled Trial of Attentional Control Training for Treating Alcohol Use Disorder
Brief Title: Attentional Control Training for Treating Alcohol Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Kjeld Andersen, Clinical professor, consultant psychiatrist, Ph.D, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 71941
Record Dates: First submitted 2021-09-18; First posted 2021-11-02 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Alcohol Use Disorder (AUD); Attentional Bias
Keywords: Cognitive bias; Attentional bias; Alcohol use disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: a gamified AACTP smartphone application + treatment as usual (TAU) (Experimental)
  Interventions: Behavioral: Attentional Control Training Program
- Group B: a gamified AACTP sham-control application + TAU (Placebo Comparator)
  Interventions: Behavioral: Attentional Control Training Program

INTERVENTIONS:
Behavioral: Attentional Control Training Program — The 268 patients fulfilling the eligibility criteria will be randomized to one of the three groups: Group A: AACTP delivered via a smartphone application + treatment as usual (TAU; n = 134), or Group B: ACTP sham training delivered via a smartphone application + TAU (n = 134) Patients in Group A will receive seven sessions of AACTP (one session per week for seven weeks). Patients in Group B will receive seven sessions of sham training (one session per week for seven weeks).

SUMMARY:
Background: There is consistent evidence that community and clinical samples of individuals with an alcohol use disorder (AUD) have attentional biases toward alcohol cues. The alcohol attentional control training program (AACTP) has shown promise for retraining these biases and decreasing alcohol consumption in community samples of excessive drinkers. However, there is a lack of evidence regarding the effectiveness of ACTP in clinical AUD samples. The main aim of the present study is to investigate whether primary pharmacological and psychological, evidence-based alcohol treatment can be enhanced by the addition of a gamified AACTP smartphone application for patients with an AUD.

Design and methods: The study will be implemented as a randomized controlled trial. A total of 268 consecutively enrolled patients with AUD will be recruited from alcohol outpatient clinics in Denmark. Patients will be randomized to one of three groups upon initiation of primary alcohol treatment: Group A: a gamified AACTP smartphone application + treatment as usual (TAU); or Group B: a gamified AACTP sham-control application + TAU. Treatment outcomes will be assessed at baseline, post-treatment, and at 3- and 6-month follow-ups. Repeated measures MANOVA will be used to compare the trajectories of the groups over time on alcohol attentional bias, alcohol craving, and drinking reductions. It is hypothesized that Group A will achieve better treatment outcomes than either Group B.

Perspectives: Because attentional bias for alcohol cues is proportional to the amount of alcohol consumed, and these biases are not addressed within current evidence-based treatment programs, this study is expected to provide new evidence regarding the effectiveness of the gamified AACTP in a clinical population. Furthermore, due to promising results found using AACTP in community samples of excessive drinkers, there is a high probability that the AACTP treatment in this study will also be effective, thereby allowing AACTP to be readily implemented in clinical settings. Finally, it is expected that this study will increase the effectiveness of evidence-based AUD treatment and introduce a new, low-cost gamified treatment targeting patients with an AUD. Overall, this study is likely to have an impact at the scientific, clinical, and societal levels.

ELIGIBILITY:
To be eligible to participate, patients must fulfill the following criteria.

Inclusion criteria:

They must (1) sign written informed consent, (2) be between 18 and 65 years old (because the intervention is web-based), (3) be fluent in Danish, (4) have completed detoxification (if deemed appropriate), (5) have been admitted to primary treatment within the past eight weeks.

Exclusion criteria:

Be color-blind, have a severe psychiatric or neurological illness (e.g., a psychotic disorder, intellectual disability, dementia) or terminal physical illness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Alcohol consumption | Baseline, post-treatment (12-weeks after baseline) and 12- and 24-weeks post-treatment follow-up
  Alcohol consumption will be measured with the Alcohol Timeline Follow-back (TLFB) method. It involves using a calendar to help the patient retrospectively recall the number of drinks that he/she consumed on each day during the previous three months. The results will be used to calculate change over time in various alcohol consumption measures, including weekly mean drinking, which will be the primary outcome measure.
  To validate the TLFB, hair samples from the patients will be tested for ethyl glucuronide (ETG) by liquid chromatography-tandem mass spectrometry (LC-MS/MS). This biological marker of alcohol consumption will be collected and analyzed according to the Society for Hair Testing.

SECONDARY OUTCOMES:
Cravings | Baseline, post-treatment (12-weeks after baseline) and 12- and 24-weeks post-treatment follow-up
  A visual analog scale (VAS) will be used to measure patients' alcohol cravings on a scale ranging from 0 to 10, with 0 indicating no craving at all and 10 indicating extreme craving. The scale will be presented visually on a ruler, and patients will be asked to indicate their mean and peak level of craving during the past 30 days.
Readiness to change | Baseline, post-treatment (12-weeks after baseline) and 12- and 24-weeks post-treatment follow-up
  The Readiness-to-Change Questionnaire Treatment Version (RTCQ-TV) is a 12-item measure of patients' stated intentions to change their drinking, which includes the following sub-scales: (1) pre-contemplation, (2) contemplation, and (3) action stages. Four items pertain to each sub-scale, and each item is rated on a 5-point Likert Scale ranging from strongly agree (-2) to strongly disagree (+2). The total score can range from -24 to +24.
Affective state | Baseline, post-treatment (12-weeks after baseline) and 12- and 24-weeks post-treatment follow-up
  The Positive and Negative Affect Schedule (PANAS) is a 20-item measure of the patient's affective states, which includes two sub-scales: (1) positive affect and (2) negative affect. Ten items pertain to each sub-scale, and each item is rated on a 5-point scale ranging from 1 (not at all) to 5 (very much). The total score can range from 20 to 100.

CONTACTS AND LOCATIONS:
Locations (1):
- KABS City, Valby, Capital Region of Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No
The datasets pertaining to the study are available on request from the authors, provided this is compliant with national legislations and with the decisions of the ethical committees of the respective countries.

REFERENCES:
- [Background] Mellentin AI, Cox WM, Fadardi JS, Martinussen L, Mistarz N, Skot L, Romer Thomsen K, Mathiasen K, Lichtenstein M, Nielsen AS. A Randomized Controlled Trial of Attentional Control Training for Treating Alcohol Use Disorder. Front Psychiatry. 2021 Nov 26;12:748848. doi: 10.3389/fpsyt.2021.748848. eCollection 2021. PMID 34899419